CLINICAL TRIAL: NCT03261531
Title: Effect of T6 Dermatome Electrical Stimulation on Gastric Motor Functions, Appetite, Satiation, Satiety and Weight Loss in Individuals With Overweight and Class I Obesity
Brief Title: Dermatome Electrical Stimulation on Individuals With Overweight and Class I Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device failure
Sponsor: Mayo Clinic (Other)
Collaborators: Elira Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-001916
Record Dates: First submitted 2017-08-08; First posted 2017-08-25 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Overweight; Class I Obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcutaneous electrical nerve stimulation (TENS) (Experimental): Healthy volunteers who are overweight or have class I obesity will receive T6 dermatomal electrical stimulation via Transcutaneous electrical nerve stimulation (TENS)
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Participants will be treated before and after two meals of the day with T6 dermatomal electrical stimulation delivered by a TENS unit.

SUMMARY:
Investigators are doing this research study to find out the effect of T6 dermatomal electrical stimulation (delivered by a Transcutaneous Electrical Nerve Stimulation (TENS) unit) on appetite and weight loss.

DETAILED DESCRIPTION:
Participants will be treated before and after two meals of the day with T6 dermatomal electrical stimulation delivered by a Transcutaneous Electrical Nerve Stimulation (TENS) unit. Participants will receive 15-minute T6 dermatome cutaneous stimulation with TENS unit applied immediately before ingestion of two of main meals of the day (breakfast and evening meal), and 60 minute stimulation applied immediately after ingestion of these meals. Participants will apply the stimulus four times daily for a treatment period of at least 3 months. Participants will keep a diary of weight once weekly and a weekly appetite record.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese adults (BMI ≥25 kg/m2 and ≤34.99 kg/m2) residing within 125 miles of Mayo Clinic in Rochester, Minnesota; these will be otherwise healthy individuals with no unstable psychiatric disease and not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine (other than hyperglycemia on diet) disorders.
* Age: 18-65 years
* Gender: Men or women. Women of childbearing potential will be using an effective form of contraception, and have negative pregnancy tests within 48 hours of enrollment and before each radiation exposure.
* Subjects must have the ability to provide informed consent before any trial-related activities.

Eligible individuals will be asked to avoid taking additional medications and supplements for the duration of the study, unless reviewed and approved by the study team.

Exclusion Criteria:

* Abdominal surgery other than appendectomy, Caesarian section or tubal ligation
* Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility, appetite or absorption, e.g., Orlistat
* Positive history of diabetes mellitus or use of hypoglycemic medications
* Positive history of spinal cord injury and/or chronic back pain
* Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD) (12), a self-administered alcoholism screening test (AUDIT-C) (13), and the Questionnaire on Eating and Weight Patterns (binge eating disorders and bulimia) (14). If such a dysfunction is identified by a HAD score >11 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Intake of medication, whether prescribed or over the counter (except multivitamins), within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, thyroxine replacement therapy, low dose analgesia or anti-inflammatory medications (Acetaminophen and Ibuprofen) and any medication administered for co-morbidities as long as they do not alter gastrointestinal motility including gastric emptying and gastric accommodation.
* Subjects may also be excluded from participation for other factors at the discretion of the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, M.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Started | 7
Completed | 3
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change in body weight will be measured in kilograms or pounds
Time Frame: Baseline, 3 months
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

2. Primary Outcome: Gastric Half-emptying Time (GE T 1/2)
Description: The time for half of the ingested solids to leave the stomach
Time Frame: After 1 day treatment (approximately at 4 hours)
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

3. Primary Outcome: Gastric Half-emptying Time (GE T 1/2)
Description: The time for half of the ingested solids to leave the stomach
Time Frame: At 3 months, approximately 2 hours after radiolabeled meal is ingested
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

4. Secondary Outcome: Fasting Gastric Volume by 99mTc-SPECT Imaging
Description: A noninvasive SPECT method will be used to measure gastric volume. Subjects will report to the clinic after an overnight fast. The first fasting scan will be obtained, and the study medication (99mTc) will be given subcutaneously. After 10 min, a 2nd fasting post medication scan will be obtained. Each scan requires about 9-12 min. Tomographic images of the gastric wall will be obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content. Volume will be measured in mL.
Time Frame: At 3 months, approx 20 minutes after 99mTC injection
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

5. Secondary Outcome: Postprandial Gastric Volume (Gastric Accommodation) by 99mTc-SPECT Imaging
Description: A noninvasive SPECT method will be used to measure gastric volume after a liquid nutritional supplement meal. Subjects reported to the clinic after an overnight fast. 99mTC will be given by an intravenous injection in the forearm. The first fasting scan was obtained, and the study medication (99mTc) will be given subcutaneously. After 10 min, a 2nd fasting post medication scan was obtained, and the meal consumed; then two serial postprandial scans will be obtained. Each scan requires about 9-12 min. Tomographic images of the gastric wall will be obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content. Volume will be measured in mL.
Time Frame: At 3 months, approximately 30 min after liquid meal
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Gastric Emptying Percentage
Description: The time for gastric retention of ingested solids or liquid to leave the stomach, measured in percentage.
Time Frame: Day 1, 3 months
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

7. Secondary Outcome: Satiation Volume (Level 3)
Description: Subjects will ingest a liquid nutrient drink at a rate of 120 mL every 4 minutes; the volume ingested at each level of fullness will be recorded. Participants record their sensations of fullness using a numerical scale from 0 to 5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal ("volume to fullness"), and level 5 corresponding to the maximum tolerated volume (MTV). Nutrient intake is stopped when subjects reach the score of 5.
Time Frame: Approximately 30 minutes after the liquid meal
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

8. Secondary Outcome: Satiation Maximum Tolerated Volume (Level 5)
Description: as for outcome 7
Time Frame: Approximately 30 minutes after the liquid meal
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Kcal Intake at Buffet Meal as a Measure of Appetite
Description: Assessment of kcal intake as a measure of appetite buffet meal to measure total caloric intake. 5 hours after ingesting 300 mL liquid nutrient as part of the gastric volume study, participants will be invited to eat, during a 30-minute period, a standard "free feeding" meal. The total amount of food consumed will be analyzed by the study dietitian.
Time Frame: At 3 months, approximately 30 minutes after the buffet meal
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Appetite Score
Description: Ratings of appetite will be measured every 30 minutes between the time of ingestion of standard liquid breakfast and the start of the ad libitum meal. The appetite rating will be measured by 4- 100 mm long Visual Analog Scales (VAS). The VAS does not have any pre-set marks between the extremes of 0 for negative rating and 100 mm for positive rating. The investigator measures the mark made by the participant in mm and records this for the value. The overall appetite score will be calculated as the average of the four individual scores (satiety + fullness+100-prospective food consumption + hunger/4.
Time Frame: Baseline, 3 months
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Fasting and Peak Postprandial Plasma Ghrelin at 3 Months
Description: Total ghrelin will be measured by a radioimmunoassay technique.
Time Frame: baseline, 90 minutes postprandially
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Fasting and Peak Postprandial Glucagon-like Peptide-1 (GLP-1) at 3 Months
Description: Glucagon-like peptide-1 (GLP-1) will be measured by a radioimmunoassay technique.
Time Frame: baseline, 90 minutes postprandially
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Fasting and Peak Postprandial Peptide Tyrosine Tyrosine (PYY) at 3 Months
Description: Peptide Tyrosine Tyrosine (PYY) will be measured by radioimmunoassay.
Time Frame: baseline, 90 minutes postprandially
Population: Study was terminated due to device failure. Sincere efforts were made but we were unable to collect data
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 3 months for each subject
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03261531/Prot_SAP_000.pdf